CLINICAL TRIAL: NCT04466150
Title: Impact of Ocrelizumab on Cerebrospinal Fluid Biomarkers at Multiple Sclerosis Onset
Acronym: IMPACT MS
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry); Valhalla Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RO-IIS-2018-10828
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Relapsing Multiple Sclerosis; Clinically Isolated Syndrome
MeSH Terms: interventions — ocrelizumab

STUDY DESIGN:
Intervention Model Description: This is a nested case-controlled study.
  By nesting this ocrelizumab interventional treatment arm within an observational study, the investigators will be able to compare treatment with ocrelizumab to usual care for patients who are matched for the same disease duration. Because the same clinical and biomarker assessments will be acquired for both the ocrelizumab interventional arm and the usual care observational cohort, this study will allow direct comparison of ocrelizumab with a usual care control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ocrelizumab treated (Active Comparator): Participants age 18-50 with a first clinical presentation of MS or high-risk CIS diagnosed within 90 days of screening will be treated with ocrelizumab (300 mg IV x 2 doses given 2 weeks apart) at disease origin and with maintenance ocrelizumab 600 mg every 6 months through 30 months with a final study visit at 3 years
  Interventions: Drug: Ocrelizumab
- Observational study cohort (No Intervention): Subjects enrolled into an observational study matched for the same disease duration and who are either untreated or treated with alternate MS disease modifying therapies will serve as a parallel reference group

INTERVENTIONS:
Drug: Ocrelizumab — open label biomarker study
  Other Names: Ocrevus
  Arms: Ocrelizumab treated

SUMMARY:
Newly diagnosed relapsing multiple sclerosis (MS) and high risk clinically isolated syndrome (CIS) patients will be treated with ocrelizumab at disease onset to see if treatment favorably alters CSF markers of chronic inflammation.

DETAILED DESCRIPTION:
Newly diagnosed relapsing multiple sclerosis (MS) and high risk clinically isolated syndrome (CIS) patients age 18-50 will be treated with ocrelizumab within 90 days of first clinical MS/CIS presentation and re-dosed as maintenance therapy every 6 months for 3 years to see if treatment favorably alters CSF markers of chronic inflammation

Investigators hope data that will provide a foundation for further studies that treating relapsing MS patients at clinical onset (using a B-cell depleting therapy) may improve longer-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria to be included in this study:

* Signed Consent Form
* High-risk clinically isolated syndrome or relapsing MS Diagnosis (based on 2017 International Panel Criteria)
* Age 18-50 inclusive
* Screening within 90 days of first clinical demyelinating event typical of MS with 1 or more inactive lesions typical of MS
* No prior MS disease modifying therapy
* No corticosteroids within 7 days of first ocrelizumab treatment
* EDSS < 4.0
* A negative urine or serum pregnancy test must be available for premenopausal women and for women <12 months after the onset of menopause, unless they have undergone surgical sterilization.
* Women of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or use one method of contraception with a failure rate of <1% per year or a barrier method supplemented with spermicide. Contraception must continue for the duration of study treatment and for at least 24 weeks after the last dose of study treatment. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause of other than menopause), and has not undergone surgical sterilization (removal of the ovaries and/or uterus).

  * Examples of contraceptive methods with a failure rate of <1% per year include bilateral tube ligation, male sterilization, established hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence and withdrawal are not acceptable methods of contraception.
  * Examples of barrier methods supplemented with the use of spermicide include male or female condom, cap, diaphragm, or sponge.

Exclusion Criteria:

Patients will be excluded from the study based on the following criteria:

* Pregnancy, lactation, or intention to become pregnant during the study
* Progressive MS (primary or secondary)
* Disease other than MS to explain the first demyelinating event; including AQP4 IgG seropositivity
* Unwilling or unsafe to proceed with CSF exams based on coagulopathy or anatomy or other considerations in the judgment of the study investigator
* Unwilling or unsafe to proceed with MRI
* Active hepatitis B virus infection
* Untreated latent or active tuberculosis
* Active hepatitis C virus infection
* HIV infection
* Hypersensitivity to trial medications
* History of life-threatening infusion reaction to MAbs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of intrathecal synthesis of gammaglobulins in treatment-naïve relapsing MS and clinically isolated syndrome participants before and after treatment with ocrelizumab | 3 years
  Comparison of intrathecal synthesis of gammaglobulins in treatment-naïve relapsing MS and clinically isolated syndrome participants before and after 3 years of treatment with ocrelizumab. Intrathecal synthesis is measured by either a) normalization of the IgG Index (0.6 is the upper limit of normal) or b) eradication of oligoclonal bands

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Cree, MD, PhD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Outcome data (biomarker, genotypic) as well as study data related to diagnosis, disease presentation, and date of birth, along with biological specimens collected as part of the study, may be shared (in coded form) in the future with other qualified researchers, government data registries, and/or commercial entities on a case by case basis at the discretion of the PI and Co-PIs. Any such investigator/entity will be required to provide appropriate documentation that the research being conducted has been approved by an Institutional Review Board and demonstrate that it will be of scientific value.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Clinical study report to Sponsor estimated May 2025. Other data/samples will be shared after initial results are published and on a case by case basis.
Access Criteria: Collaborators, other scientific Investigators, Government Health and research agencies, Commercial Companies may request data and/or samples. The request process includes submitting a research proposal, having necessary IRB approval and material transfer agreements.

REFERENCES:
- [Background] Lassmann H, Bradl M. Multiple sclerosis: experimental models and reality. Acta Neuropathol. 2017 Feb;133(2):223-244. doi: 10.1007/s00401-016-1631-4. Epub 2016 Oct 20. PMID 27766432
- [Background] Bruck W, Gold R, Lund BT, Oreja-Guevara C, Prat A, Spencer CM, Steinman L, Tintore M, Vollmer TL, Weber MS, Weiner LP, Ziemssen T, Zamvil SS. Therapeutic decisions in multiple sclerosis: moving beyond efficacy. JAMA Neurol. 2013 Oct;70(10):1315-24. doi: 10.1001/jamaneurol.2013.3510. PMID 23921521
- [Background] Longbrake EE, Cross AH. Effect of Multiple Sclerosis Disease-Modifying Therapies on B Cells and Humoral Immunity. JAMA Neurol. 2016 Feb;73(2):219-25. doi: 10.1001/jamaneurol.2015.3977. PMID 26720195
- [Background] van Oosten BW, Lai M, Hodgkinson S, Barkhof F, Miller DH, Moseley IF, Thompson AJ, Rudge P, McDougall A, McLeod JG, Ader HJ, Polman CH. Treatment of multiple sclerosis with the monoclonal anti-CD4 antibody cM-T412: results of a randomized, double-blind, placebo-controlled, MR-monitored phase II trial. Neurology. 1997 Aug;49(2):351-7. doi: 10.1212/wnl.49.2.351. PMID 9270561
- [Background] Li R, Rezk A, Miyazaki Y, Hilgenberg E, Touil H, Shen P, Moore CS, Michel L, Althekair F, Rajasekharan S, Gommerman JL, Prat A, Fillatreau S, Bar-Or A; Canadian B cells in MS Team. Proinflammatory GM-CSF-producing B cells in multiple sclerosis and B cell depletion therapy. Sci Transl Med. 2015 Oct 21;7(310):310ra166. doi: 10.1126/scitranslmed.aab4176. PMID 26491076
- [Background] Dobson R, Ramagopalan S, Davis A, Giovannoni G. Cerebrospinal fluid oligoclonal bands in multiple sclerosis and clinically isolated syndromes: a meta-analysis of prevalence, prognosis and effect of latitude. J Neurol Neurosurg Psychiatry. 2013 Aug;84(8):909-14. doi: 10.1136/jnnp-2012-304695. Epub 2013 Feb 21. PMID 23431079
- [Background] Howell OW, Reeves CA, Nicholas R, Carassiti D, Radotra B, Gentleman SM, Serafini B, Aloisi F, Roncaroli F, Magliozzi R, Reynolds R. Meningeal inflammation is widespread and linked to cortical pathology in multiple sclerosis. Brain. 2011 Sep;134(Pt 9):2755-71. doi: 10.1093/brain/awr182. Epub 2011 Aug 11. PMID 21840891
- [Background] Magliozzi R, Howell OW, Reeves C, Roncaroli F, Nicholas R, Serafini B, Aloisi F, Reynolds R. A Gradient of neuronal loss and meningeal inflammation in multiple sclerosis. Ann Neurol. 2010 Oct;68(4):477-93. doi: 10.1002/ana.22230. PMID 20976767
- [Background] Stashenko P, Nadler LM, Hardy R, Schlossman SF. Characterization of a human B lymphocyte-specific antigen. J Immunol. 1980 Oct;125(4):1678-85. PMID 6157744
- [Background] Krumbholz M, Derfuss T, Hohlfeld R, Meinl E. B cells and antibodies in multiple sclerosis pathogenesis and therapy. Nat Rev Neurol. 2012 Nov 5;8(11):613-23. doi: 10.1038/nrneurol.2012.203. Epub 2012 Oct 9. PMID 23045237
- [Background] Leandro MJ, Cambridge G, Ehrenstein MR, Edwards JC. Reconstitution of peripheral blood B cells after depletion with rituximab in patients with rheumatoid arthritis. Arthritis Rheum. 2006 Feb;54(2):613-20. doi: 10.1002/art.21617. PMID 16447239
- [Background] Salzer J, Svenningsson R, Alping P, Novakova L, Bjorck A, Fink K, Islam-Jakobsson P, Malmestrom C, Axelsson M, Vagberg M, Sundstrom P, Lycke J, Piehl F, Svenningsson A. Rituximab in multiple sclerosis: A retrospective observational study on safety and efficacy. Neurology. 2016 Nov 15;87(20):2074-2081. doi: 10.1212/WNL.0000000000003331. Epub 2016 Oct 19. PMID 27760868
- [Background] Chamberlain N, Massad C, Oe T, Cantaert T, Herold KC, Meffre E. Rituximab does not reset defective early B cell tolerance checkpoints. J Clin Invest. 2016 Jan;126(1):282-7. doi: 10.1172/JCI83840. Epub 2015 Dec 7. PMID 26642366
- [Background] Cree BA, Lamb S, Morgan K, Chen A, Waubant E, Genain C. An open label study of the effects of rituximab in neuromyelitis optica. Neurology. 2005 Apr 12;64(7):1270-2. doi: 10.1212/01.WNL.0000159399.81861.D5. PMID 15824362
- [Background] Hauser SL, Waubant E, Arnold DL, Vollmer T, Antel J, Fox RJ, Bar-Or A, Panzara M, Sarkar N, Agarwal S, Langer-Gould A, Smith CH; HERMES Trial Group. B-cell depletion with rituximab in relapsing-remitting multiple sclerosis. N Engl J Med. 2008 Feb 14;358(7):676-88. doi: 10.1056/NEJMoa0706383. PMID 18272891
- [Background] Bar-Or A, Calabresi PA, Arnold D, Markowitz C, Shafer S, Kasper LH, Waubant E, Gazda S, Fox RJ, Panzara M, Sarkar N, Agarwal S, Smith CH. Rituximab in relapsing-remitting multiple sclerosis: a 72-week, open-label, phase I trial. Ann Neurol. 2008 Mar;63(3):395-400. doi: 10.1002/ana.21363. PMID 18383069
- [Background] Ruhstaller TW, Amsler U, Cerny T. Rituximab: active treatment of central nervous system involvement by non-Hodgkin's lymphoma? Ann Oncol. 2000 Mar;11(3):374-5. doi: 10.1023/a:1008371602708. No abstract available. PMID 10811510
- [Background] Naismith RT, Piccio L, Lyons JA, Lauber J, Tutlam NT, Parks BJ, Trinkaus K, Song SK, Cross AH. Rituximab add-on therapy for breakthrough relapsing multiple sclerosis: a 52-week phase II trial. Neurology. 2010 Jun 8;74(23):1860-7. doi: 10.1212/WNL.0b013e3181e24373. PMID 20530322
- [Background] Alping P, Frisell T, Novakova L, Islam-Jakobsson P, Salzer J, Bjorck A, Axelsson M, Malmestrom C, Fink K, Lycke J, Svenningsson A, Piehl F. Rituximab versus fingolimod after natalizumab in multiple sclerosis patients. Ann Neurol. 2016 Jun;79(6):950-8. doi: 10.1002/ana.24651. Epub 2016 Apr 20. PMID 27038238
- [Background] Rommer PS, Dorner T, Freivogel K, Haas J, Kieseier BC, Kumpfel T, Paul F, Proft F, Schulze-Koops H, Schmidt E, Wiendl H, Ziemann U, Zettl UK; GRAID investigators. Safety and Clinical Outcomes of Rituximab Treatment in Patients with Multiple Sclerosis and Neuromyelitis Optica: Experience from a National Online Registry (GRAID). J Neuroimmune Pharmacol. 2016 Mar;11(1):1-8. doi: 10.1007/s11481-015-9646-5. Epub 2015 Nov 20. PMID 26589235
- [Background] Hauser SL, Bar-Or A, Comi G, Giovannoni G, Hartung HP, Hemmer B, Lublin F, Montalban X, Rammohan KW, Selmaj K, Traboulsee A, Wolinsky JS, Arnold DL, Klingelschmitt G, Masterman D, Fontoura P, Belachew S, Chin P, Mairon N, Garren H, Kappos L; OPERA I and OPERA II Clinical Investigators. Ocrelizumab versus Interferon Beta-1a in Relapsing Multiple Sclerosis. N Engl J Med. 2017 Jan 19;376(3):221-234. doi: 10.1056/NEJMoa1601277. Epub 2016 Dec 21. PMID 28002679
- [Background] Klein C, Lammens A, Schafer W, Georges G, Schwaiger M, Mossner E, Hopfner KP, Umana P, Niederfellner G. Epitope interactions of monoclonal antibodies targeting CD20 and their relationship to functional properties. MAbs. 2013 Jan-Feb;5(1):22-33. doi: 10.4161/mabs.22771. Epub 2012 Dec 4. PMID 23211638
- [Background] Kappos L, Li D, Calabresi PA, O'Connor P, Bar-Or A, Barkhof F, Yin M, Leppert D, Glanzman R, Tinbergen J, Hauser SL. Ocrelizumab in relapsing-remitting multiple sclerosis: a phase 2, randomised, placebo-controlled, multicentre trial. Lancet. 2011 Nov 19;378(9805):1779-87. doi: 10.1016/S0140-6736(11)61649-8. Epub 2011 Oct 31. PMID 22047971
- [Background] Sorensen PS, Lisby S, Grove R, Derosier F, Shackelford S, Havrdova E, Drulovic J, Filippi M. Safety and efficacy of ofatumumab in relapsing-remitting multiple sclerosis: a phase 2 study. Neurology. 2014 Feb 18;82(7):573-81. doi: 10.1212/WNL.0000000000000125. Epub 2014 Jan 22. PMID 24453078
- [Background] Bar-Or A, Grove RA, Austin DJ, Tolson JM, VanMeter SA, Lewis EW, Derosier FJ, Lopez MC, Kavanagh ST, Miller AE, Sorensen PS. Subcutaneous ofatumumab in patients with relapsing-remitting multiple sclerosis: The MIRROR study. Neurology. 2018 May 15;90(20):e1805-e1814. doi: 10.1212/WNL.0000000000005516. Epub 2018 Apr 25. PMID 29695594
- [Background] Weinshenker BG, Bass B, Rice GP, Noseworthy J, Carriere W, Baskerville J, Ebers GC. The natural history of multiple sclerosis: a geographically based study. I. Clinical course and disability. Brain. 1989 Feb;112 ( Pt 1):133-46. doi: 10.1093/brain/112.1.133. PMID 2917275
- [Background] Tremlett H, Zhao Y, Devonshire V; UBC Neurologists. Natural history comparisons of primary and secondary progressive multiple sclerosis reveals differences and similarities. J Neurol. 2009 Mar;256(3):374-81. doi: 10.1007/s00415-009-0039-7. Epub 2009 Mar 18. PMID 19308306
- [Background] Confavreux C, Vukusic S, Moreau T, Adeleine P. Relapses and progression of disability in multiple sclerosis. N Engl J Med. 2000 Nov 16;343(20):1430-8. doi: 10.1056/NEJM200011163432001. PMID 11078767
- [Background] Polman CH, Reingold SC, Banwell B, Clanet M, Cohen JA, Filippi M, Fujihara K, Havrdova E, Hutchinson M, Kappos L, Lublin FD, Montalban X, O'Connor P, Sandberg-Wollheim M, Thompson AJ, Waubant E, Weinshenker B, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2010 revisions to the McDonald criteria. Ann Neurol. 2011 Feb;69(2):292-302. doi: 10.1002/ana.22366. PMID 21387374
- [Background] Ontaneda D, Thompson AJ, Fox RJ, Cohen JA. Progressive multiple sclerosis: prospects for disease therapy, repair, and restoration of function. Lancet. 2017 Apr 1;389(10076):1357-1366. doi: 10.1016/S0140-6736(16)31320-4. Epub 2016 Nov 24. PMID 27889191
- [Background] Hawker K, O'Connor P, Freedman MS, Calabresi PA, Antel J, Simon J, Hauser S, Waubant E, Vollmer T, Panitch H, Zhang J, Chin P, Smith CH; OLYMPUS trial group. Rituximab in patients with primary progressive multiple sclerosis: results of a randomized double-blind placebo-controlled multicenter trial. Ann Neurol. 2009 Oct;66(4):460-71. doi: 10.1002/ana.21867. PMID 19847908
- [Background] Montalban X, Hauser SL, Kappos L, Arnold DL, Bar-Or A, Comi G, de Seze J, Giovannoni G, Hartung HP, Hemmer B, Lublin F, Rammohan KW, Selmaj K, Traboulsee A, Sauter A, Masterman D, Fontoura P, Belachew S, Garren H, Mairon N, Chin P, Wolinsky JS; ORATORIO Clinical Investigators. Ocrelizumab versus Placebo in Primary Progressive Multiple Sclerosis. N Engl J Med. 2017 Jan 19;376(3):209-220. doi: 10.1056/NEJMoa1606468. Epub 2016 Dec 21. PMID 28002688
- [Background] Dyson JK, Jopson L, Ng S, Lowery M, Harwood J, Waugh S, Valappil M, McPherson S. Improving testing for hepatitis B before treatment with rituximab. Eur J Gastroenterol Hepatol. 2016 Oct;28(10):1172-8. doi: 10.1097/MEG.0000000000000689. PMID 27388147
- [Background] Lee J, Park JY, Huh KH, Kim BS, Kim MS, Kim SI, Ahn SH, Kim YS. Rituximab and hepatitis B reactivation in HBsAg-negative/anti-HBc-positive kidney transplant recipients. Nephrol Dial Transplant. 2017 May 1;32(5):906. doi: 10.1093/ndt/gfx048. No abstract available. PMID 28371939
- [Background] Seto WK, Wong DK, Chan TS, Hwang YY, Fung J, Liu KS, Gill H, Lam YF, Cheung KS, Lie AK, Lai CL, Kwong YL, Yuen MF. Association of Hepatitis B Core-Related Antigen With Hepatitis B Virus Reactivation in Occult Viral Carriers Undergoing High-Risk Immunosuppressive Therapy. Am J Gastroenterol. 2016 Dec;111(12):1788-1795. doi: 10.1038/ajg.2016.436. Epub 2016 Sep 20. PMID 27644733
- [Background] Clifford DB, Ances B, Costello C, Rosen-Schmidt S, Andersson M, Parks D, Perry A, Yerra R, Schmidt R, Alvarez E, Tyler KL. Rituximab-associated progressive multifocal leukoencephalopathy in rheumatoid arthritis. Arch Neurol. 2011 Sep;68(9):1156-64. doi: 10.1001/archneurol.2011.103. Epub 2011 May 9. PMID 21555606
- [Background] Hauser SL. The Charcot Lecture | beating MS: a story of B cells, with twists and turns. Mult Scler. 2015 Jan;21(1):8-21. doi: 10.1177/1352458514561911. Epub 2014 Dec 5. PMID 25480864
- [Background] Harding K, Williams O, Willis M, Hrastelj J, Rimmer A, Joseph F, Tomassini V, Wardle M, Pickersgill T, Robertson N, Tallantyre E. Clinical Outcomes of Escalation vs Early Intensive Disease-Modifying Therapy in Patients With Multiple Sclerosis. JAMA Neurol. 2019 May 1;76(5):536-541. doi: 10.1001/jamaneurol.2018.4905. PMID 30776055
- [Background] Brown JWL, Coles A, Horakova D, Havrdova E, Izquierdo G, Prat A, Girard M, Duquette P, Trojano M, Lugaresi A, Bergamaschi R, Grammond P, Alroughani R, Hupperts R, McCombe P, Van Pesch V, Sola P, Ferraro D, Grand'Maison F, Terzi M, Lechner-Scott J, Flechter S, Slee M, Shaygannejad V, Pucci E, Granella F, Jokubaitis V, Willis M, Rice C, Scolding N, Wilkins A, Pearson OR, Ziemssen T, Hutchinson M, Harding K, Jones J, McGuigan C, Butzkueven H, Kalincik T, Robertson N; MSBase Study Group. Association of Initial Disease-Modifying Therapy With Later Conversion to Secondary Progressive Multiple Sclerosis. JAMA. 2019 Jan 15;321(2):175-187. doi: 10.1001/jama.2018.20588. PMID 30644981
- [Background] Ontaneda D, Tallantyre EC, Raza PC, Planchon SM, Nakamura K, Miller D, Hersh C, Craner M, Bale C, Chaudhry B, Gunzler DD, Love TE, Gerry S, Coles A, Cohen JA, Evangelou N. Determining the effectiveness of early intensive versus escalation approaches for the treatment of relapsing-remitting multiple sclerosis: The DELIVER-MS study protocol. Contemp Clin Trials. 2020 Aug;95:106009. doi: 10.1016/j.cct.2020.106009. Epub 2020 Apr 19. PMID 32320842
- [Background] raditional Versus Early Aggressive Therapy for Multiple Sclerosis Trial (TREAT-MS) Johns Hopkins University NCT03500328
- [Background] University of California, San Francisco MS-EPIC Team; Cree BAC, Hollenbach JA, Bove R, Kirkish G, Sacco S, Caverzasi E, Bischof A, Gundel T, Zhu AH, Papinutto N, Stern WA, Bevan C, Romeo A, Goodin DS, Gelfand JM, Graves J, Green AJ, Wilson MR, Zamvil SS, Zhao C, Gomez R, Ragan NR, Rush GQ, Barba P, Santaniello A, Baranzini SE, Oksenberg JR, Henry RG, Hauser SL. Silent progression in disease activity-free relapsing multiple sclerosis. Ann Neurol. 2019 May;85(5):653-666. doi: 10.1002/ana.25463. Epub 2019 Mar 30. PMID 30851128
- [Background] Warnke C, Stettner M, Lehmensiek V, Dehmel T, Mausberg AK, von Geldern G, Gold R, Kumpfel T, Hohlfeld R, Maurer M, Stangel M, Straeten V, Limmroth V, Weber T, Kleinschnitz C, Wattjes MP, Svenningsson A, Olsson T, Hartung HP, Hermsen D, Tumani H, Adams O, Kieseier BC. Natalizumab exerts a suppressive effect on surrogates of B cell function in blood and CSF. Mult Scler. 2015 Jul;21(8):1036-44. doi: 10.1177/1352458514556296. Epub 2014 Nov 12. PMID 25392339
- [Background] Larsson D, Akerfeldt T, Carlson K, Burman J. Intrathecal immunoglobulins and neurofilament light after autologous haematopoietic stem cell transplantation for multiple sclerosis. Mult Scler. 2020 Oct;26(11):1351-1359. doi: 10.1177/1352458519863983. Epub 2019 Jul 26. PMID 31347948
- [Background] Rejdak K, Stelmasiak Z, Grieb P. Cladribine induces long lasting oligoclonal bands disappearance in relapsing multiple sclerosis patients: 10-year observational study. Mult Scler Relat Disord. 2019 Jan;27:117-120. doi: 10.1016/j.msard.2018.10.006. Epub 2018 Oct 10. PMID 30368223
- [Background] Leist TP, Comi G, Cree BA, Coyle PK, Freedman MS, Hartung HP, Vermersch P, Casset-Semanaz F, Scaramozza M; oral cladribine for early MS (ORACLE MS) Study Group. Effect of oral cladribine on time to conversion to clinically definite multiple sclerosis in patients with a first demyelinating event (ORACLE MS): a phase 3 randomised trial. Lancet Neurol. 2014 Mar;13(3):257-67. doi: 10.1016/S1474-4422(14)70005-5. Epub 2014 Feb 4. PMID 24502830
- [Background] https://www.emdserono.com/content/dam/web/corporate/non-images/country-specifics/us/pi/mavenclad-pi.pdf
- [Background] https://www.gene.com/download/pdf/ocrevus_prescribing.pdf.